CLINICAL TRIAL: NCT02479269
Title: The Influence of Aerobic Exercise on Serum Brain Natriuretic Peptide and C- Reactive Protein in Cardiovascular Disease
Acronym: AEBNPCRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Islamic Azad University, Shiraz (Other)
Responsible Party: Principal Investigator, Najmeh Sheykhiyan, Master, Islamic Azad University, Shiraz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CT-P-92-6517
Record Dates: First submitted 2015-06-13; First posted 2015-06-24 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Cardiovascular Disease
Keywords: Brain Natriuretic Peptide; aerobic execise; C- Reactive Protein
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention (Experimental): Aerobic exercise+ blood sampling
  Interventions: Other: Aerobic exercise
- control (No Intervention): Blood sampling

INTERVENTIONS:
Other: Aerobic exercise — Aerobic exercise for 8 weeks
  Arms: intervention

SUMMARY:
The purpose of this study was to investigate the effects of 8 weeks of aerobic exercise on serum concentrations of Brain Natriuretic Peptide and C - reactive protein in patients with cardiovascular disease. Patients were divided randomly into two groups: control and experimental aerobic group. This study was done with two - stage blood sampling: at the beginning and at the end of the treatment phase. All subjects were requested to avoid any exercise at least 48 hours before blood sampling. To study Brain Natriuretic Peptide and C - reactive protein changes, 5 milliliters of blood were taken from patient's brachial vein. Blood samples for subsequent measurements were frozen immediately and transported to the Hormone Laboratory for serum separation. The experimental group did the aerobic exercise programs for 8 weeks for 3 sessions per week and the control group did not receive any training. After completion of training, the final blood samplings were performed. Exercise intensity according to the heart rate remained stable until the last week. Brain Natriuretic Peptide and C - reactive protein levels were measured by ELISA tests. All statistical analysis were done using SPSS software (version 16) and at the significance level of p≤ 0.05

ELIGIBILITY:
Inclusion Criteria:

* In this trial patients with coronary artery disease more than 70 percent at least in one coronary vessel with Ejection Fraction more than 40 percent in recent Echo cardiograph without acute evidence of ischemia or congestive heart failure symptoms were selected and are divide randomly into two groups.

Exclusion Criteria:

* Patients with acute evidence of ischemia or congestive heart failure symptoms are excluded.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Brain Natriuretic Peptide | 8 weeks
serum C - reactive protein | 8 weeks

SECONDARY OUTCOMES:
serum lipoproteins | 8 weeks
Body Mass Index | 8 weeks
blood pressure | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mohammad Ali Ostovan, Cardiologist, Study Director — Shiraz University of Medical Sciences